CLINICAL TRIAL: NCT06698809
Title: Obstructive Sleep Apnea Therapeutic Intervention for REsiDual Sleepiness (STILL TIRED)
Brief Title: Obstructive Sleep Apnea Therapeutic Intervention for REsiDual Sleepiness
Acronym: STIL TIRED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-00907
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea; Sleepiness
Keywords: Transcranial Photobiomodulation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleepiness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Participants with Moderate-to-Severe OSA (Experimental): Participants will receive tPBM treatment and sham for approximately 12 minutes and complete assessments. Participants have the choice to participate in an optional follow-up 1 week post-initial visit, in which they will receive tPBM treatment for approximately 11-12 minutes and complete assessments at a different time of day.
  Interventions: Device: Active tPBM

INTERVENTIONS:
Device: Active tPBM — tPBM is a neuromodulatory treatment that uses red and/or near infrared light to penetrate the cortex and can alter both cerebral metabolism and blood flow. Subjects will receive treatment for approximately 12 minutes per treatment and sham.

SUMMARY:
Obstructive sleep apnea (OSA) is a sleep disorder that is commonly treated using positive airway pressure, yet 50% of patients still experience residual sleepiness after successful therapy. A potential neuromodulation strategy that can decrease residual sleepiness is transcranial photobiomodulation (tPBM). tPBM is a neuromodulatory treatment that uses red and/or near infrared light to penetrate the cortex and can alter both cerebral metabolism and blood flow. However, this potential has never been explored before directly in sleep disordered individuals. This project aims to explore the effect of tPBM on sleepiness and understand the potential neural mechanism of tPBM in OSA. The short-term goal of this project is to collect pilot data, which is the first of its kind, and suggest tPBM as a potential modulator of sleepiness in OSA.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively normal (Telephone Interview for Cognitive Status (TiCS) ≥29))
* Moderate - severe OSA
* Currently on therapy for OSA and has received treatment for OSA for at least 3 months.
* Sustained compliance with continuous positive airway pressure (CPAP), which means using the machine at least 4 hours per night for five nights a week.
* Epworth Sleepiness Score (ESS) greater than or equal to 8 or excess daytime sleepiness as defined by the Functional Outcome Sleep Questionnaire or clinical complaint.

Exclusion Criteria:

* Documented diagnosis of chronic insomnia, or sleep onset insomnia based on Insomnia Severity Index (ISI)
* Documented diagnosis of circadian rhythm disorder
* Any current use of supplemental oxygen
* Other sleep-related breathing disorders (central sleep apnea, etc.) based on American Academy of Sleep Medicine (AASM) criteria
* Current shift work involving night shift (regular work between 12am and 6am or night shift) within the past 6 months
* Anticipated scheduled bariatric surgery within the next 3 months
* Chronic regular (> 2 nights per week) use of any sedative, stimulant, neuroleptic drugs, or other medications limiting validity of cognitive tests. This includes regular use of alcohol or marijuana for sleep. Melatonin is ok.
* Diagnosis of uncontrolled psychiatric disease in the last six months, and/or history of schizophrenia or bipolar disorder. Controlled conditions will include major depressive disorder, panic disorder, schizoaffective disorder, generalized anxiety disorder, Obsessive-compulsive disorder (OCD), substance use disorders, and alcohol abuse/dependence. Personality disorders and neurodevelopmental disorders (e.g. autism, ADHD) are allowed if cognition is within normal limits.
* Taking methylphenidate for ADHD.
* Presence of other critical comorbid conditions that would lead to inability to complete the study protocol (including follow-up for 2 years), or that would affect cognition (e.g. clinically relevant endocrine or hematological conditions).
* Chronic regular (> 2 nights per week) use of stimulant if unable to complete a washout prior to MRI.
* Does not have a regular sleeping environment (i.e., sleeps in a different setting > 2 nights per week).
* Currently pregnant or planning to become pregnant.
* Prior diagnosis of a Central nervous system (CNS) disease, such as multiple sclerosis, stroke, Parkinson's disease, Alzheimer's disease, epilepsy, a loss of consciousness > 24 hours, or traumatic brain injury as identified by the Cumulative Illness Rating Scale for Geriatrics (CIRS). Participants who are diagnosed with Mild cognitive impairment (MCI) or Alzheimer's disease based on neuropsychological testing will be excluded. Delirium in the last 12 months.
* Near-miss or prior automobile accident "due to sleepiness" within the past 12 months.
* Employed as a commercial driver during the study (for example, bus drivers, train engineers, airplane pilots) or construction worker.
* Past intolerance or hypersensitivity to tPBM.
* Significant skin conditions (i.e., hemangioma, scleroderma, psoriasis, rash, open wound or tattoo) on the subject's scalp that are found in the area of the procedure sites.
* Any use of light-activated drugs (photodynamic therapy) within 14 days prior to study enrollment.
* Any type of implants in the head, whose functioning might be affected by tPBM (e.g., stent, clipped aneurysm, embolized arteriovenous malformation (AVM), implantable shunt - Hakim valve).
* Failure to meet standard MRI safety requirements (e.g., claustrophobia, non-removable piercings, implanted medical devices, other non-removable metals) as determined by the MRI Safety Checklist.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-03 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Cerebral Blood Flow | Pre-Active tPBM Treatment, Post-Active tPBM Treatment (Day 1, approx. 11-12 minutes)
  Measured via MRI imaging.

SECONDARY OUTCOMES:
Change in Karolinska Sleepiness Scale (KSS) Score | Pre-Active tPBM Treatment, Post-Active tPBM Treatment (Day 1, approx. 11-12 minutes)
  The KSS is a 1-item assessment of sleepiness in the 5 minutes prior to administration of the questionnaire. Participants rank their sleepiness on a scale from 1 (extremely alert) to 9 (very sleepy). The total score is the item ranking and ranges from 1-9; higher scores indicate greater sleepiness.
Change in Psychomotor Vigilance Task (PVT) Score | Pre-Active tPBM Treatment, Post-Active tPBM Treatment (Day 1, approx. 11-12 minutes)
  The psychomotor vigilance task (PVT) is a computer-based test that measures how consistently someone responds to visual or auditory stimuli over 10 minutes. The participant presses a button in response to a digital signal on a computer screen. The test measures reaction time and the number of lapses, which are defined as response times longer than 500 milliseconds or failing to respond. The total score is calculated by subtracting the number of lapses and false starts from 100%. The result is a percentage that ranges from 100% for optimal performance to 0% for worst possible performance.
Change in Controlled Oral Word Association Test (COWAT) Score | Pre-Active tPBM Treatment, Post-Active tPBM Treatment (Day 1, approx. 11-12 minutes)
  The COWAT is a verbal fluency test in which participants are asked to say as many words as possible from a given category and in a specified timeframe. The total score is the number of correct words named by the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Gaggi, Principal Investigator — NYU Langone Health; Ricardo Osario, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Naomi.Gaggi@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Naomi.Gaggi@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.